CLINICAL TRIAL: NCT02867085
Title: A Prospective Longitudinal Cohort Study to Investigate the Interactions of Bone and Hematopoiesis in the Elderly
Brief Title: Study Investigating the Interactions of Bone and Hematopoiesis in the Elderly
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: BoHemE
Record Dates: First submitted 2016-07-27; First posted 2016-08-15 (Estimated); Last update posted 2025-08-24 (Actual); Status verified 2024-11

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS; Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Group 1 (MDS group)
  Interventions: Other: Observational
- Group 2 (control group)
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — The BoHemE study does not provide any recommendations for treatment. Guidelines for osteoporosis treatment and standardized instructions for MDS patients are available, however the choice of treatment is up to the treating physician and should be reported as such.

SUMMARY:
The prospective BoHemE study is designed to evaluate the correlation between bone marrow function and skeletal health in elderly patients (>= 60 years) with or without pre-existing myelodysplastic syndromes (MDS).

ELIGIBILITY:
Inclusion Criteria Group 1 (MDS group):

* Age ≥60 years
* With known or suspected MDS (according WHO, <20% blast count)
* Written informed consent

Inclusion Criteria Group 2 (control group):

* Age ≥60 years
* Undergoing elective knee or hip replacement therapy
* Normal blood count (defined by Hb ♀ >12 g/dL, ♂ >13 g/dL; ANC >1.8x10^9/L; PLT >100x10^9/L)
* Written informed consent

Exclusion Criteria Group 1 (MDS group) + 2 (control group):

* History of bilateral total hip replacement prior to study
* Control group only: diagnosis of MDS or AML prior to study
* Dementia defined as MMSE score of <24
* Renal insufficiency with an eGFR <30 mL/min
* Liver cirrhosis Child-Pugh B or C
* Active infection (HIV, hepatitis B or C, tuberculosis)
* Heart insufficiency NYHA III or IV or severe cardiac valve disease
* Prior allogeneic stem cell transplantation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The BoHemE study includes elderly patients (≥60 years) with or without MDS and age-related concomitant diseases.
  The therapeutic management of patients is subject to current treatment recommendations and is determined solely by the attending physician. It is planned to include at least 356 patients (i. e. 178 per group) exhibiting the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
T score of bone mineral density at the total hip and at lumbar spine L1-L4 in elderly patients with MDS and a control group without MDS. Osteoporosis is defined as a T score of <-2.5 at the hip and at lumbar spine L1-L4. | five years

SECONDARY OUTCOMES:
Time-dependent molecular patterns of clonality and their association with secondary malignancies and outcome in healthy and MDS individuals | five years
  Composite measures as part of a patient registry
Hematological profile of MDS patients (karyotype, immunophenotype, molecular characteristics, WHO and IPSS R classification, therapy) | five years
  Composite measures as part of a patient registry
Sociodemographic parameters (age, sex, socioeconomic status) | five years
  Composite measures as part of a patient registry
Disease characteristics (onset/date of diagnosis of MDS and osteoporosis, previous treatments and diagnostic results) | five years
  Composite measures as part of a patient registry
Clinical osteoporotic fractures | five years
Quality of life (QLQ C30, SF 36) | five years
  Composite measures as part of a patient registry
Medical care (Number of medical consultations/hospital admissions due to osteoporosis, medical professions, falls) | five years
  Composite measures as part of a patient registry
Comorbidities (Hematopoietic Cell Transplantation-specific Comorbidity Index) | five years
Disease evolution of MDS (change of MDS subtype according to IPSS-R and WHO classification) | five years
  Composite measures as part of a patient registry
Disease evolution of osteoporosis (measured by number of fractures within the previous 24 months) | five years
Overall survival | five years
  Duration from the day of study entry to the day of death

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Platzbecker, MD, Principal Investigator — Universität Leipzig; Lorenz C. Hofbauer, MD, Principal Investigator — Technische Universität Dresden
Locations (2):
- Germany (2):
  - Universitätsklinikum Dresden, Dresden
  - Universitätsklinikum Leipzig, Leipzig

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schneider M, Rolfs C, Trumpp M, Winter S, Fischer L, Richter M, Menger V, Nenoff K, Grieb N, Metzeler KH, Kubasch AS, Sockel K, Thiede C, Wu J, Woo J, Bruderle A, Hofbauer LC, Lutzner J, Roth A, Cross M, Platzbecker U. Activation of distinct inflammatory pathways in subgroups of LR-MDS. Leukemia. 2023 Aug;37(8):1709-1718. doi: 10.1038/s41375-023-01949-2. Epub 2023 Jul 7. PMID 37420006